CLINICAL TRIAL: NCT01566227
Title: Within-subject Comparison of Mandibular Overdentures Retained by 1,2,or 3 Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, IPesun (1), Department Head, Restorative Dentistry Department, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: B2012:012
Record Dates: First submitted 2012-02-20; First posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Complete Edentulism
Keywords: overdenture; implant; edentulism
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- number of implants (Experimental): number of implants (1,2 or 3) used to retained an overdenture
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — 3 surveys with 10 questions each: one before, during and after treatment
  Other Names: Satisfaction survey; questionnaire for patient satisfaction

SUMMARY:
This research is being done to find out the ideal number of implants/attachments required to provide adequate stability of dentures during function.

DETAILED DESCRIPTION:
The aim of this study is threefold: i) to evaluate within-subject response to complete lower dentures retained by 1 or 2 or 3 implants fitted with independent overdenture attachments; ii) laboratory evaluation of the retention force generated with 1-2 or 3-implants and study its correlation to patients' response; iii) study the wear pattern of the plastic inserts on the overdenture abutments during each retention mode (i.e. the number of implants used to retain the dentures) and correlate its effects to denture stability.

ELIGIBILITY:
Inclusion Criteria:

* subjects completely edentulous on maxilla and mandible for at least a year (w/out dentures)
* Adult age (25 plus) male or female
* Stable medical health
* Ability to participate in the study for at least 3-4 years
* Able to understand and respond to surveys used in the study
* Adequate amount of bone in the mandible to receive 3 implants.

Exclusion Criteria:

history of drug and alcohol abuse, excessive smoking (more than 1 pack/day)

* surgical limitations:
* uncontrolled systemic disease: diabetes, etc.. that may compromised healing
* irradiated surgical site
* inadequate bone height and width (re: implant size)
* inability to undergo minor oral surgery because of health or personal reasons
* psychological and handicapped conditions that may hinder 4-year involvement (physical handicap conditions)
* Severe TMDs related to joint pathology

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction survey (questionnaires) | every 6 months up to three years
  Assess efficacy of treatment by analysis of patient's answer to a satisfaction survey.

SECONDARY OUTCOMES:
Radiographs | every 6 months up to three years
  Assess crestal bone level around the implants.
Wear of 1 vs 2 vs 3 GPS retention components on complete dentures. | baseline and 6 months
  The force required to remove the female retentive componenets from the male component will be compaired between one vs two vs three retentive components.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Pesun, DDS, Principal Investigator — Univ. of Manitoba, Faculty of Dentistry; Reynaldo Todescan, DDS., Study Director — Univ of Manitoba, Faculty of Dentistry; Mike Barczac, DDS, Study Chair — Univ of Manitoba, Faculty of Dentistry
Locations (1):
- University of Manitoba, Faculty of Dentistry, Winnipeg, Manitoba, Canada